CLINICAL TRIAL: NCT06558240
Title: To Explore the Effectiveness and Feasibility of HERADERM Hydrogel Wound Dressing on Caesarean Section Surgical Site
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chia-Hao Liu, Visiting Staff, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2024-08-023AC
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-08

CONDITIONS: Cesarean Section; Surgical Wound; Surgical Wound Infection; Wounds and Injuries
Keywords: cesarean section; wound healing; HERADERM Hydrogel Wound Dressing (Sterile); surgical site infection; wound care
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection; Wounds and Injuries; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: HERADERM Hydrogel Wound Dressing (Sterile): Eligible subjects will use experimental dressings for postoperative wound care after caesarean section. The subjects received dressing change on the second day after surgery and on the day of discharge. After discharge, subjects will take home 2 pieces of experimental dressings and change by themselves.
  (Timing to change dressing after discharge: the area of exudate exceeds two-thirds of the dressing area)
  Interventions: Device: HERADERM Hydrogel Wound Dressing (Sterile)

INTERVENTIONS:
Device: HERADERM Hydrogel Wound Dressing (Sterile) — HERADERM Hydrogel Wound Dressing (Sterile) is a transparent, composite hydrogel dressing. The outer layer is a waterproof and breathable polyurethane film (PU film), which can prevent external bacterial invasion and reduce the risk of infection. The inner layer is A+ polymer hydrogel, which can keep the wound bed in a moist state and reduce the infiltration problem caused by wound exudate.

SUMMARY:
The wound of cesarean section involves multiple layers of tissue and often cause significant postoperative pain. The epidermal wound typically heals within 1 to 2 weeks after surgery. In current clinical practice, advanced wound dressings are commonly used for postoperative wound care. The theory of moist wound healing was first proposed by Winter in 1962, advocating that maintaining a moist environment around the wound can accelerate the healing process.

HERADERM Hydrogel Wound Dressing (Sterile) was approved by the Taiwan FDA in 1999. Although HERADERM Hydrogel Wound Dressing (Sterile) are frequently used clinically for post-cesarean section wound care, there have been no comprehensive reports evaluating the effectiveness and clinical application of the dressings to date. The purpose of this study is to explore the effectiveness and feasibility of HERADERM Hydrogel Wound Dressing on caesarean section surgical site and to provide user experience and clinical data for reference by patients and clinical personnel.

DETAILED DESCRIPTION:
In this observational, prospective, single-arm study. We aimed to explore the effectiveness and feasibility of HERADERM Hydrogel Wound Dressing (Sterile) on caesarean section surgical site. Written informed consent are obtained before subjects participate in the study. Eligible subjects will be taken initial wound photos and use experimental dressings for postoperative wound care after closure of caesarean section wound site. To evaluate the clinical applicability of the experimental dressings, wound healing assessments will be conducted by independent study nurse during the postoperative period, hospitalization, and follow-up visits. Information of pain intensity experienced by subjects during dressing removal will be collected. Additionally, satisfaction surveys based on subjects' experiences of wearing and changing the experimental dressings will also be collected during the hospitalization and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18, scheduling for a transverse incision cesarean section, and using HERADERM Hydrogel Wound Dressing (Sterile) for wound care at the end of the surgery.
2. Gestational age over 37 weeks on the day of the cesarean section.
3. Body mass index (BMI) less than 35 kg/m² on the day of the cesarean section.
4. Subjects must be able to comply with follow-up wound care visits and subsequent monitoring.

Exclusion Criteria:

1. Subjects unwilling to sign the consent form or with poor compliance.
2. Currently suffering from severe immune-related skin diseases, such as severe urticaria, generalized eczema, pemphigus, lupus erythematosus, etc.
3. Using medications that affect wound healing (e.g., glucocorticoids, anticoagulants and immunosuppressive drugs).
4. Subjects were deemed unsuitable for participation by investigator, such as uncontrolled infection and conditions that interfere with wound healing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects going to undergo cesarean section
Study Population: Subjects going to have cesarean section in Taipei Veterans General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
REEDA scale | Assessing on post-operative day 2, 4 & 11
  The scale includes five factors that indicate abdominal wound healing: redness, edema, ecchymosis, discharge, and approaching wound edges. Each improvement factor is evaluated by giving 0, 1, 2 and 3 points. The sum of the scores obtained as a result of the evaluation of five categories constitutes the REEDA score. The lowest score on the scale is 0, and the highest score is 15. The highest score on the scale indicates severe perineal trauma.
Percentage of surgical wound infection | Assessing on post-operative day 2, 4 & 11 if there are any surgical site infection
  The definition of surgical site infection will be according to CDC definitions of nosocomial surgical site infections: a modification of CDC definitions of surgical wound infection.

SECONDARY OUTCOMES:
Percentage of allergic reaction to experimental dressings | Within 11 days after surgery
  The incidence of allergic reaction related to the experimental dressings will be recorded. The final wound check will be performed by the surgeon at 11 days postoperatively.
Intensity of pain during dressing removal | Assessing on post-operative day 2, 4 & 11
  Pain intensity is assessed by Numerical Rating Scale (NRS). Numerical Rating Scale was a 11-point scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Incidence of adverse events | Within 11 days after surgery
  The incidence of postoperative adverse events related to the experimental dressings will be recorded.
Number of dressing change | Within 11 days after surgery
  Subjects will take home 2 pieces of experimental dressings and change by themselves. Number of dressing change will be recorded at 11 days postoperatively.
Satisfaction survey | Assessing on post-operative day 2, 4 & 11
  Subjects' and caregivers' satisfaction survey regarding user experience quantified with the use of a 5-grade scale with 'highly satisfied', 'satisfied', 'uncertain', 'dissatisfied' or 'very dissatisfied'.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hao Liu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No